CLINICAL TRIAL: NCT05525637
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Phase 3 Clinical Study to Evaluate the Efficacy and Safety of YZJ-1139 Tablets in the Treatment of Insomnia Disorder
Brief Title: Safety and Efficacy Study of YZJ-1139 in Insomnia Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YZJ-1139-3-01
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YZJ-1139 20mg (Experimental)
  Interventions: Drug: YZJ-1139 20mg
- YZJ-1139 40mg (Experimental)
  Interventions: Drug: YZJ-1139 40mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YZJ-1139 20mg — YZJ-1139 20mg tablets, once daily in the evening
  Arms: YZJ-1139 20mg
Drug: YZJ-1139 40mg — YZJ-1139 40mg tablets, once daily in the evening
  Arms: YZJ-1139 40mg
Drug: Placebo — Match placebo tablets, once daily in the evening
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess efficacy and safety of YZJ-1139 in adult subjects with insomnia disorder. Efficacy will be evaluated on objective and subjective sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

- Subjects who meet all of the following criteria may be enrolled in the study:

1. Aged ≥ 18 to < 65 years.
2. Meet the clinical diagnostic criteria for insomnia disorder as defined in International Classification of Sleep Disorders, 3rd Edition (ICSD-3) criteria.
3. sTSO ≥ 30 min for at least 3 nights per week and/or sWASO ≥ 60 min for at least 3 nights per week within 28 days (4 weeks) prior to screening.
4. During the run-in period or on Day 1 of the treatment period, sTSO ≥ 30 min for at least 3 nights in the last 7 sleep diaries and/or sWASO ≥ 60 min for at least 3 nights out of 7 nights as confirmed by the sleep diary prior to Polysomnography (PSG) monitoring.
5. PSG results for 2 consecutive nights during the run-in period should meet the following conditions:

   * The mean LPS of 2 nights is ≥ 30 min, with the LPS ≥ 20 min for any night;
   * And/or the mean WASO of 2 nights is ≥ 60 min, with neither night < 45 min;
   * The mean SE of 2 nights is ≤ 85%, with the SE ≤ 87.5% for both nights.
6. ISI score ≥ 15 at screening and on Day 1 of the treatment period.
7. Agree to follow the habitual bedtime between 9 p.m. and 1 a.m., wake up between 5 a.m. and 10 a.m. every day, and stay in bed for 6.5 to 9 hours per night during the study.
8. Have a bedtime between 9 p.m. and 1 a.m., wake up between 5 a.m. and 10 a.m., and stay in bed for 6.5 to 9 hours for at least 5 days in the last 7 sleep diaries as confirmed by the sleep diary prior to PSG monitoring during the run-in period or on Day 1 of the treatment period.
9. Female subjects are confirmed to be non-pregnant at screening; both men of reproductive potential and women of childbearing potential should agree to use medically acceptable and effective contraception throughout the study and within 3 months after the end of the study.
10. Understand the study procedures and contents, voluntarily participate in the clinical study and sign the written Informed Consent Form (ICF), have good compliance during participation in the study, and are willing to attend the visits.

Exclusion Criteria:

* Subjects who meet any of the following criteria should be excluded from this study:

  1. Depression: Hamilton Depression Scale (HAMD) score ≥ 18; anxiety: Hamilton Anxiety Scale (HAMA) score ≥ 14.
  2. Suicidal ideation with or without plan at screening or within 6 months prior to screening (score ≥ 3 on item 3 [suicide] of HAMD, or select "Yes" on item 3, 4 or 5 of suicidal ideation subscale of Columbia-Suicide Severity Rating Scale (C-SSRS)), or have any suicidal behavior in the past 10 years (as assessed by the suicidal ideation subscale of C-SSRS).
  3. Apnea-hypopnea index (AHI) and/or periodic limb movement index (PLMI) > 10 times/hour detected by PSG monitoring during the run-in period.
  4. Repeat electrocardiogram (ECG) at screening shows QTcF interval prolongation (QTcF > 450 ms) (the ECG should be repeated 2 more times only if the initial ECG shows QTcF interval > 450 ms).
  5. Have serious endocrine diseases, hematological diseases, cardiovascular and cerebrovascular diseases, gastrointestinal diseases, liver and kidney diseases, autoimmune diseases, impaired respiratory function or other related diseases, or have other medical history that may affect the safety of the subjects or interfere with the study assessments in the opinion of the investigator.
  6. Have insomnia disorder due to other causes such as chronic pain, headache, eczema, neurodermatitis, allergic rhinitis, and serious dermatitis (difficulty sleeping due to physical reasons, difficulty falling asleep due to medical reasons).
  7. Previous history of nervous system disorders such as epilepsy, schizophrenia, bipolar mental disorder, neurodevelopmental retardation, and cognitive disorder, or previous history of other mental illness that may affect the safety of the subjects or interfere with the study assessments in the opinion of the investigator.
  8. Previous history of sleep-related respiratory disorders including obstructive sleep apnea (with or without continuous positive airway pressure (CPAP) therapy), periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disturbances, narcolepsy or other sleep disorders: subjects with restless legs syndrome which is diagnosed by relevant diagnostic and treatment guidelines should be excluded.
  9. Have previous complex sleep behaviors, such as sleep driving, sleep eating, and sleep phone calls.
  10. Plan to undergo surgery during the study.
  11. Have received any hypnotics, antidepressants, antipsychotic drugs, anticholinergics, memory-enhancing drugs, antihistamines, centrally acting analgesics, centrally acting muscle relaxants, central nervous system stimulants, cytochrome P450 3A (CYP3A) inducers, CYP3A inhibitors, traditional Chinese medicines and traditional Chinese medicinal products with sleep-improving effects, or any other therapies for insomnia disorder within 1 week prior to the run-in period or within 5 half-lives of the investigational product, whichever is longer.
  12. History of drug taking or addiction, which is known through questioning.
  13. Have any lifestyle that interferes with the study process or may interfere with sleep: for example, there will be travels across 3 or more time zones (mainland China is considered as 1 time zone) within the next 2 weeks or during the study period, or there will be shift work (night and daytime shift).
  14. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2 × the upper limit of normal (ULN), or Creatinine (Cr) > 1.5 × ULN.
  15. Hyperthyroidism.
  16. History of alcohol abuse (defined as regular daily alcohol consumption exceeding the following criteria: approximately 720 mL of beer, or 240 mL of wine, or 60 mL of liquor) within the past 2 years.
  17. History of drug abuse within the past 2 years, or positive urine drug screening for any indicator.
  18. Regular daily consumption of excessive tea and coffee drinks (defined as consumption of > 4 cups of caffeinated beverages or > 400 mg of caffeine per day), or daily habituation to drinking caffeinated beverages beyond 18:00.
  19. Have nocturia increased caused by urinary tract infection, urinary tract injury or prostatic disorder.
  20. Have positive infectious disease screening for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb) and human immunodeficiency virus (HIV) antibody at screening.
  21. Unable to avoid vaccination within 1 month prior to screening or during the first treatment phase.
  22. Have participated in clinical studies of other drugs within the past 1 month or 5 half-lives (whichever is longer), or plan to participate in other studies simultaneously during participation in this study.
  23. Pregnant or lactating women.
  24. History of allergy to the investigational product or its components.
  25. Have prior participation in clinical studies of YZJ-1139 Tablets.
  26. Have other conditions that make the subject unsuitable for participation in the clinical study in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1041 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the subjective sleep efficiency (sSE) after 14 days of treatment | from baseline to week 2
  Subjective Sleep efficiency variation assessed by the sleep diary questionnaire at 14 days of treatment from baseline. A positive change from baseline indicates an increase in the subjective Sleep efficiency. A negative change from baseline indicates a decrease in subjective Sleep efficiency
Change from baseline in the sleep efficiency (SE) after 14 days of treatment | from baseline to day 14
  Sleep efficiency variation assessed by polysomnography at 14 days of treatment from baseline. A positive change from baseline indicates an increase in the Sleep efficiency. A negative change from baseline indicates a decrease in Sleep efficiency

SECONDARY OUTCOMES:
Change from baseline in the subjective sleep efficiency (sSE) after 7 days of treatment | Baseline, week 1
  sSE is self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the Subjective time to sleep onset (sTSO) after 14 days of treatment for subjects entering the second treatment phase | Baseline, week 1, week 2
  sTSO are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the Subjective wake after sleep onset (sWASO) after 14 days of treatment for subjects entering the second treatment phase | Baseline, week 1, week 2
  sWASO are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the Subjective total sleep time (sTST) after 14 days of treatment for subjects entering the second treatment phase | Baseline, week 1, week 2
  sTST are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the Subjective number of awakenings (sNAW) after 14 days of treatment for subjects entering the second treatment phase | Baseline, week 1, week 2
  sNAW are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the SE after 2 days of treatment | Baseline, Day1/Day2
  SE assessed by polysomnography at 2 days of treatment from baseline. A positive change from baseline indicates an increase in the Sleep efficiency. A negative change from baseline indicates a decrease in Sleep efficiency
Latency to persistent sleep (LPS) after 2 and 14 days of treatment | Baseline, Day1/Day2, Day13/Day14
  LPS assessed by polysomnography at 2 and 14 days of treatment from baseline. A positive change from baseline indicates an increase in the Sleep efficiency. A negative change from baseline indicates a decrease in Sleep efficiency
Wake after sleep onset (WASO) after 2 and 14 days of treatment | Baseline, Day1/Day2, Day13/Day14
  WASO assessed by polysomnography at 2 and 14 days of treatment from baseline. A positive change from baseline indicates an increase in the Sleep efficiency. A negative change from baseline indicates a decrease in Sleep efficiency
Total sleep time (TST) after 2 and 14 days of treatment | Baseline, Day1/Day2, Day13/Day14
  TST assessed by polysomnography at 2 and 14 days of treatment from baseline. A positive change from baseline indicates an increase in the Sleep efficiency. A negative change from baseline indicates a decrease in Sleep efficiency
Sleep structure (wakefulness, N1, N2, N3, rapid eye movement sleep [REM], non-rapid eye movement sleep [NREM], REM latency, number of awakenings [NAW], arousal index for REM and NREM) after 2 and 14 days of treatment | Baseline, Day1/Day2, Day13/Day14
  Sleep structure assessed by polysomnography at 2 and 14 days of treatment from baseline.
Change from baseline in the mean subjective sleep quality score after 7 and 14 days of treatment for subjects | Baseline, Week 1, Week 2
  Subjective sleep quality score is a self-report assessment of participant perception of the effects of a medication on their sleep. Higher score indicated severe insomnia problem.
Percentage of Participants on each scale of Global Impression of Insomnia (PGI-I) each Item at 14 days of treatment | Day 14
  The PGI-I was a self-report assessment of participant perception of the effects of a medication on their sleep. The PGI-I had 3 items related to study medication effects (a) helped/worsened sleep, (b) decreased/increased time to fall asleep, (c) increased/decreased total sleep time, and 1 item related to perceived appropriateness of study medication strength. The first 3 items were answered on a 3-point scale (1=positive medication effect, 2=neutral medication effect, 3=negative medication effect) and the last item on a different 3 point scale (medication: 1=too strong, 2=just right, 3=too weak)
Changes from baseline in the sSE after 30, 90 and 180 days of treatment for subjects entering the second treatment phase | Baseline, Day 30, Day 90, and Day 180
  sSE are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the sTSO after 30, 90 and 180 days of treatment for subjects entering the second treatment phase | Baseline, Day 30, Day 90, and Day 180
  sTSO are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the sWASO after 30, 90 and 180 days of treatment for subjects entering the second treatment phase | Baseline, Day 30, Day 90, and Day 180
  sWASO are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the sTST after 30, 90 and 180 days of treatment for subjects entering the second treatment phase | Baseline, Day 30, Day 90, and Day 180
  sTST are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Changes from baseline in the sNAW after 30, 90 and 180 days of treatment for subjects entering the second treatment phase | Baseline, Day 30, Day 90, and Day 180
  sNAW are self-reported sleep outcome measured by subject diary data, collected daily and analyzed at appropriate intervals.
Change from baseline in the mean subjective sleep quality score after 30, 90 and 180 days of treatment for subjects entering the second treatment phase | Baseline, Day 30, Day 90, and Day 180
  Subjective sleep quality score is a self-report assessment of participant perception of the effects of a medication on their sleep. Higher score indicated severe insomnia problem.
Change from baseline in the Insomnia Severity Index (ISI) score after 30, 90 and 180 days of treatment for subjects entering the second treatment phase | Baseline, Day 30, Day 90, and Day 180
  ISI is a self-report questionnaire assessing the nature, severity, and impact of insomnia. Higher score indicated severe insomnia problem.
Percentage of Participants who enter the second treatment phase on each scale of Patient Global Impressions - ImprovementGlobal Impression of Insomnia (PGI-I) each Item at 30, 90 and 180 days of treatment | Day 30, Day 90, and Day 180
  The PGI-I was a self-report assessment of participant perception of the effects of a medication on their sleep. The PGI-I had 3 items related to study medication effects (a) helped/worsened sleep, (b) decreased/increased time to fall asleep, (c) increased/decreased total sleep time, and 1 item related to perceived appropriateness of study medication strength. The first 3 items were answered on a 3-point scale (1=positive medication effect, 2=neutral medication effect, 3=negative medication effect) and the last item on a different 3 point scale (medication: 1=too strong, 2=just right, 3=too weak).

CONTACTS AND LOCATIONS:
Locations (88):
- China (88):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Beijing Hui Long Guan Hospital, Capital Medical University, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First affiliated hospital of bengbu medical college, Bengbu
  - Binzhou Medical University Hospital, Binzhou
  - The First Bethune Hospital Of Jilin University, Changchun
  - The First Hospital of ChangSha, Changsha
  - The Second XiangYa Hospital Of Central University, Changsha
  - The Secong People's Hospital Of HuNan Province, Changsha
  - Xiangya Hospital Central South University, Changsha
  - ChengDu Second People's Hospital, Chengdu
  - The Fourth People's Hospital Of ChengDu, Chengdu
  - Army Medical Center of PLA, Chongqing
  - ChongQing Eleventh People's Hospital, Chongqing
  - ChongQing Mental Health Center, Chongqing
  - ChongQing Traditional Chinese Medical Hospital, Chongqing
  - ChongQing University Three Gorges Hospital, Chongqing
  - People's Hospital Of DeYang City, Deyang
  - The First Affiliated Hospital Of FuJan Medical University, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Nanfang Hospital Southern Medical University, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - The Affiliated Hospital Of GuiZhou Medical University, Guiyang
  - HanDan Central Hospital, Handan
  - Affiliated HangZhou First People's Hospital, Hangzhou
  - Sir Run Run Shaw hospital, Hangzhou
  - The 2nd Affiliated Hospital Of Harbin Medical University, Ha’erbin
  - Chaohu hospital of anhui medical university, Hefei
  - The Second Hospital Of AnHui Medical University, Hefei
  - The Secong People's Hospital Of HeFei, Hefei
  - Affiliated NanHua Hospital,University Of South China, Hengyang
  - JiangMen Central Hospital, Jiangmen
  - ShanDong Provincial QianFoShan Hospital, Jinan
  - Jingjiang People's Hospital, Jingjiang
  - Shandong Daizhuang Hospital, Jining
  - Jiujiang University Affiliated Hospital, Jiujiang
  - First People's Hospital of Yunnan Province, Kunming
  - LiaoCheng People's Hospital, Liaocheng
  - HeNan University Of Science &Technology, Luoyang
  - The Affiliated Hospital Of Southwest Medical University, Luzhou
  - JiangXi Provincial People's Hospital, Nanchang
  - The First Affiliated Hospital Of NanChang University, Nanchang
  - The Second Affiliated Hospital Of NanChang University, Nanchang
  - NanJing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast Unveristy, Nanjing
  - NanTong First People's Hospital, Nantong
  - NingBo KangNing Hospital, Ningbo
  - NingBo Medical Center LiHuiLi Hospital, Ningbo
  - QingDao Center Medical Group, Qingdao
  - QingDao Municipal Hospital, Qingdao
  - The affilated hospital of qingdao university, Qingdao
  - The 2nd Affiliated Hospital Of FuJan Medical University, Quanzhou
  - Affiliated ZhongShan Hospital,University Of FuDan, Shanghai
  - HuaShan Hospital Fudan University, Shanghai
  - ShangHai University Of Traditional Chinese Medical Shuguang Hospital, Shanghai
  - ShengJing Hospital Of China Medical University, Shenyang
  - ShenZhen People's Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - Jilin Neuropsychiatric Hospital, Siping
  - SuZhou GuangJi Hospital, Suzhou
  - The First People's Hospital Of KunShan, Suzhou
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - First Hospital Of ShanXi Medical University, Taiyuan
  - Peking University BinHai Hospital, Tianjin
  - Tianjin Huanhu Hospital, Tianjin
  - Tianjin Mental Health Center, Tianjin
  - The Center Hospital of WuHan, Wuhan
  - Unidn Hospital TongJi Medical College HuaZhong University Of Science And Technology, Wuhan
  - Wuhan Mental Health Centre, Wuhan
  - Affiliated Hospital Of Jiangnan University, Wuxi
  - WuXi People's Hospital, Wuxi
  - Air Force Medical University, Xi'an
  - XianYang Hospital OF Yan'an University, Xianyang
  - HeNan Mental Hospital, Xinxiang
  - The Affiliated Hospital Of XuZhou Medical University, Xuzhou
  - XuZhou Central Hospital, Xuzhou
  - HeNan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital Of ZhenZhou University, Zhengzhou
  - ZhenZhou Central Hospital, Zhengzhou
  - ZhenJiang Mental Health Center, Zhenjiang
  - ZhuMaDian Second People's Hospital, Zhumadian
  - ZiGong First People's Hospital, Zigong